CLINICAL TRIAL: NCT05913869
Title: Use of a Telehealth Approach to Build Resilience in Parents of Children With Autism Through Mindfulness Practice
Brief Title: Online Mindfulness-based Program for Parents of Children With Autism
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: San Jose State University (Other)
Responsible Party: Principal Investigator, Megan Chang, Associate professor, San Jose State University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 22124
Record Dates: First submitted 2022-09-02; First posted 2023-06-22 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-02

CONDITIONS: Mindfulness; Psychophysiologic Reaction; Behavior, Health
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Online MBSR 1 (Experimental): received modified online 8-week group-based MBSR intervention delivered by a UMASS trained MBSR instructor
  Interventions: Behavioral: Online Mindfulness Based Stress Reduction
- Waitlist control (Active Comparator): On a waiting list to receive the identical intervention as the treatment group after the active treatment group completes.
  Interventions: Behavioral: Online Mindfulness Based Stress Reduction

INTERVENTIONS:
Behavioral: Online Mindfulness Based Stress Reduction — Based on the UMASS curriculum developed by Dr. Jon Kabat-Zinn, it is an 8-week mindfulness stress reduction program. It is a skill-based psychoeducational program that meets 2 hours for 8 weeks to discuss stress, cognition and health. The weekly intervention includes didactic presentations, class dialogue and inquiry, formal (e.g., body scan, walking meditation) and informal (e.g., awareness of pleasant and unpleasant events, interpersonal communications, etc.) mindfulness practice.
  Other Names: MBSR

SUMMARY:
The goal of the project is to investigate the effects of online 8-week MBSR intervention on diverse parents to support their children with ASD. The investigators will conduct a randomized waitlist-controlled trial with a sample size 22 parents. This study utilizes psychological, behavioral and psychophysiological measures with parents of children with ASD ages 6-12. The first aim is to determine if parents of children with autism from diverse populations are willing participate in and complete an online MBSR program and if online delivery is as effective as in-person program. The battery of parental-report psychological assessments to measure resilience, parental sleep and stress as well as children's behaviors will be administered before and after the treatment. The second aim is to investigate the effects of a virtual MBSR intervention on cardiovascular and sympathetic nervous activity measured by continuous EDA and EKG. Participants will participate in a validated laboratory stress protocol consisting of mental arithmetic and speech tasks before and after the MBSR intervention.

DETAILED DESCRIPTION:
After the participants eligibility are confirmed, their signatures will be obtained on the consent form. Three data collection phases are included in this protocol: baseline, post 3 months and post 6 months. All tests are identical in which phase. Each test includes a survey packet and the lab experiment. The surveys packet includes: the Connor-Davidson Resilience Scale, Mindfulness Attention Awareness Scale, Parenting Stress Index - 4th edition Short Form, Pittsburgh Sleep Quality Index, Adult Sensory Processing Scale, Strength and Difficulties Questionnaire, and WHO Quality of Life-BREF. For the lab experiment, EKG and EDA data will be collected through lab protocol, which include a 5-min baseline recording followed by Trier Social Stress Test (speaking, math test) and then another 5-min rest period. After that, a pre-recorded 15-min mindfulness practice will be played for the participants to practice. After completing the baseline test, participants will be randomly grouped into the MBSR group or the waitlist controlled group. The online MBSR program is a 8-week group-based, intervention, which will be delivered by a UMASS trained MBSR instructor.

ELIGIBILITY:
Inclusion Criteria:

* have a child aged 6-12 years old that has been diagnosed by a psychiatrist or a psychologist with autism spectrum disorder
* English speaking
* parents do not receive any form of psychological or behavioral treatment at the time of referral
* parents have never participated in a MBSR workshop prior to the enrollment
* parents do not have previous meditation experience
* parents do not have a severe mental illness (self-assessed),
* parents agree to participate in the 8-week MBSR intervention

Exclusion Criteria:

* parents who currently receive psychotherapy or take medications for health issues

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Connor-Davidson Resilience Scale from baseline to midpoint | from baseline to midpoint (approximately 3 months from baseline)
  This standardized assessment is comprised of 25 items, which measures 7 aspects of resilience including: hardiness, coping, adaptability, self-efficacy, meaningfulness/purpose, optimism, and regulation of emotion and cognition. Each item is rated on a 5-point Likert scale. The total score ranges from zero to 100. Higher score indicate greater resilience. It has been shown to have the sensitivity to detect the treatment effects.
Change in Connor-Davidson Resilience Scale from baseline to exit evaluation | from baseline to exit evaluation (approximately 6 months from baseline)
  This standardized assessment is comprised of 25 items, which measures 7 aspects of resilience including: hardiness, coping, adaptability, self-efficacy, meaningfulness/purpose, optimism, and regulation of emotion and cognition. Each item is rated on a 5-point Likert scale. The total score ranges from zero to 100. Higher score indicate greater resilience. It has been shown to have the sensitivity to detect the treatment effects.
Change in Connor-Davidson Resilience Scale from midpoint to exit evaluation | from midpoint to exit evaluation (approximately 3 months from baseline to 6 months from baseline)
  This standardized assessment is comprised of 25 items, which measures 7 aspects of resilience including: hardiness, coping, adaptability, self-efficacy, meaningfulness/purpose, optimism, and regulation of emotion and cognition. Each item is rated on a 5-point Likert scale. The total score ranges from zero to 100. Higher score indicate greater resilience. It has been shown to have the sensitivity to detect the treatment effects.

SECONDARY OUTCOMES:
Mindfulness Attention Awareness Scale | from baseline to midpoint (approximately 3 months from baseline)
  This 15-item standardized assessment evaluates awareness of or attention to the present moment in daily life. Each item is rated on a 6-point Likert scale. The total score ranges from 15 to 90 and higher scores indicate a greater mindfulness state. Each It has moderate to strong correlations with other measures of mindfulness and has been used with families with children with ASD .
Mindfulness Attention Awareness Scale | from baseline to exit evaluation (approximately 6 months from baseline)
  This 15-item standardized assessment evaluates awareness of or attention to the present moment in daily life. Each item is rated on a 6-point Likert scale. The total score ranges from 15 to 90 and higher scores indicate a greater mindfulness state. Each It has moderate to strong correlations with other measures of mindfulness and has been used with families with children with ASD .
Mindfulness Attention Awareness Scale | from midpoint to exit evaluation (approximately 3 months from baseline to 6 months from baseline)
  This 15-item standardized assessment evaluates awareness of or attention to the present moment in daily life. Each item is rated on a 6-point Likert scale. The total score ranges from 15 to 90 and higher scores indicate a greater mindfulness state. Each It has moderate to strong correlations with other measures of mindfulness and has been used with families with children with ASD .
Parenting Stress Index - 4th edition Short Form | from baseline to midpoint (approximately 3 months from baseline)
  This index has 36 items assessing parenting-related stress that includes a Total Stress scale along with three subscales: Parental Distress, Parent-Child Dysfunctional Interaction and Difficult Child. Each item is rated on the agreement from 1= strongly agree to 5=strongly disagree. The higher scores indicate a greater perceived stress.
Parenting Stress Index - 4th edition Short Form | from baseline to exit evaluation (approximately 6 months from baseline)
  This index has 36 items assessing parenting-related stress that includes a Total Stress scale along with three subscales: Parental Distress, Parent-Child Dysfunctional Interaction and Difficult Child. Each item is rated on the agreement from 1= strongly agree to 5=strongly disagree. The higher scores indicate a greater perceived stress.
Parenting Stress Index - 4th edition Short Form | from midpoint to exit evaluation (approximately 3 months from baseline to 6 months from baseline)
  This index has 36 items assessing parenting-related stress that includes a Total Stress scale along with three subscales: Parental Distress, Parent-Child Dysfunctional Interaction and Difficult Child. Each item is rated on the agreement from 1= strongly agree to 5=strongly disagree. The higher scores indicate a greater perceived stress.
Pittsburgh Sleep Quality Index (Buysse et al., 1989) | from baseline to midpoint (approximately 3 months from baseline)
  This 19-item questionnaire measures sleep quality and quantity based on 7 components: subjective sleep quality, sleep latency, sleep duration, sleep disturbance, use of sleep medication, and daytime dysfunction and global score. The score ranges from 0 to 21 and the higher scores indicate more sleep problems
Pittsburgh Sleep Quality Index (Buysse et al., 1989) | from baseline to exit evaluation (approximately 6 months from baseline)
  This 19-item questionnaire measures sleep quality and quantity based on 7 components: subjective sleep quality, sleep latency, sleep duration, sleep disturbance, use of sleep medication, and daytime dysfunction and global score. The score ranges from 0 to 21 and the higher scores indicate more sleep problems
Pittsburgh Sleep Quality Index (Buysse et al., 1989) | from midpoint to exit evaluation (approximately 3 months from baseline to 6 months from baseline)
  This 19-item questionnaire measures sleep quality and quantity based on 7 components: subjective sleep quality, sleep latency, sleep duration, sleep disturbance, use of sleep medication, and daytime dysfunction and global score. The score ranges from 0 to 21 and the higher scores indicate more sleep problems
World Health Organization Quality of Life- BREF | from baseline to midpoint (approximately 3 months from baseline)
  This 26-item standardized questionnaire assess quality of life. It is composed of 4 domains: physical health, psychological health, social relationships, and environmental. facets. Each item is rated on a 5-point response scale and the scores are transformed linearly to a 0-100 scale. The higher score indicates higher quality of life.
World Health Organization Quality of Life- BREF | from baseline to exit evaluation (approximately 6 months from baseline)
  This 26-item standardized questionnaire assess quality of life. It is composed of 4 domains: physical health, psychological health, social relationships, and environmental. facets. Each item is rated on a 5-point response scale and the scores are transformed linearly to a 0-100 scale. The higher score indicates higher quality of life.
World Health Organization Quality of Life- BREF | from midpoint to exit evaluation (approximately 3 months from baseline to 6 months from baseline)
  This 26-item standardized questionnaire assess quality of life. It is composed of 4 domains: physical health, psychological health, social relationships, and environmental. facets. Each item is rated on a 5-point response scale and the scores are transformed linearly to a 0-100 scale. The higher score indicates higher quality of life.
Electrodermal activity (EDA) | from baseline to midpoint (approximately 3 months from baseline)
  EDA is also known as skin conductance. Two electrodes are attached to the palm to record skin conductance level that measures sweat gland activity with a sampling rate of 1000 Hz through a lab protocol. The unit of EDA is denoted as uS or microsiemens.
Electrodermal activity (EDA) | from baseline to exit evaluation (approximately 6 months from baseline)
  EDA is also known as skin conductance. Two electrodes are attached to the palm to record skin conductance level that measures sweat gland activity with a sampling rate of 1000 Hz through a lab protocol. The unit of EDA is denoted as uS or microsiemens.
Electrodermal activity (EDA) | from midpoint to exit evaluation (approximately 3 months from baseline to 6 months from baseline)
  EDA is also known as skin conductance. Two electrodes are attached to the palm to record skin conductance level that measures sweat gland activity with a sampling rate of 1000 Hz through a lab protocol. The unit of EDA is denoted as uS or microsiemens.
heart rate | from baseline to midpoint (approximately 3 months from baseline)
  continuous data recording of electrocardiogram through a lab protocol. The recording data will be processed to generate analytical data showing average heart rate per 5 minutes.
heart rate | from baseline to exit evaluation (approximately 6 months from baseline)
  continuous data recording of electrocardiogram through a lab protocol. The recording data will be processed to generate analytical data showing average heart rate per 5 minutes.
heart rate | from midpoint to exit evaluation (approximately 3 months from baseline to 6 months from baseline)
  continuous data recording of electrocardiogram through a lab protocol. The recording data will be processed to generate analytical data showing average heart rate per 5 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Megan Chang, PhD, Principal Investigator — San Jose State University
Locations (1):
- San Jose State University, San Jose, California, United States

IPD SHARING:
Plan to Share IPD: No